CLINICAL TRIAL: NCT02638922
Title: Evaluation of 304 Danish Girls With Tall Stature: Phenotypic Characteristics and Effects of Oral Administration of Natural 17β-Estradiol
Brief Title: Evaluation and Treatment of Tall Statured Girls
Acronym: TallgirlsDK
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Juul, Professor, Rigshospitalet, Denmark
Other Study IDs: RH-2015-218-04161
Record Dates: First submitted 2015-12-13; First posted 2015-12-23 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Constitutional Tall Stature
MeSH Terms: interventions — Estradiol; Trisequens

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- no treatment: girls who never received estradiol treatment
- Estradiol treatment: girls who received estradiol treatment
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol — Estradiol containing compounds administered orally in a non-randomized manner.
  Other Names: Estradiol (Trisekvens®, Novo Nordisk, Denmark),; Estradiol (Trisekvens Forte®, Novo Nordisk, Denmark); Estradiol (Femanest®, Sandoz A/S, Denmark)
  Groups: Estradiol treatment

SUMMARY:
Objective

To evaluate the phenotypic characteristics and diagnoses in a large cohort of 304 consecutive girls referred due to tall stature. Furthermore, to evaluate the effect of oral administration of 17β-estradiol on predicted adult height in constitutionally tall statured girls.

Design

A single-centre retrospective observational study of 304 girls evaluated due to tall stature between 1993 and 2013.

Setting

Tertiary referral centre for pediatric endocrinology.

Participants

A total of 304 girls were evaluated for tall stature of whom 39 (13%) were excluded due to missing data, reclassification, overgrowth syndromes or associated comorbidities. Another 58 (19%) girls did not fulfil auxological criteria for constitutionally tall stature (CTS), resulting in a total of 207 (68%) girls eligible for analysis.

Main Outcome Measures

The effect of oral treatment with 17β-estradiol on height, predicted adult height (PAH), final height and circulating hormones in constitutional tall statured girls.

DETAILED DESCRIPTION:
17α-ethinylestradiol (EE2) treatment of extreme tall stature has become increasingly debated and controversial. In Sweden, percutaneous epiphysiodesis operation is suggested as an alternative to EE2 treatment. An alternative clinical practise was introduced 20 years ago, when early treatment with oral administration of natural estrogens (17β-estradiol (E2)) was introduced in order to initiate or ensure rapid progression of puberty (and epiphyseal closure) in tall statured girls.

A retrospective 20-year single center experience included evaluation of 304 tall statured girls and the possible clinical effects of oral administration of E2.

Subjects and methods

Patients

The patient population consisted of girls who were referred with tall stature or overgrowth syndromes (ICD10 34.4, and ICD10 DE874, DQ970, DQ873A, DQ873B) to the Department of Growth and Reproduction at Rigshospitalet in Copenhagen, Denmark, during a 20-years period (between 1993 and 2013). A total of 304 patients were identified, and the diagnoses were re-evaluated as part of the present study.

Clinical data and medical history

Medical history was obtained using a structured review of patient record files. Clinical data on pubertal development were obtained from each patient visit. Puberty was evaluated by inspection and palpation of the breasts and s pubic hair according to Marshall and Tanner. A wall-mounted stadiometer (Holtain Ltd., Crymych, United Kingdom) was used to measure standing height to the nearest 0.1 cm. The girls were weighed on a digital electronic scale (Seca delta, model 707; Seca, Hamburg, Germany) with a precision of 0.1 kg while wearing light clothing and no shoes. BMI was calculated as weight (kg) divided by height (m2). The Danish growth references published by Tinggaard et al. was used in this study. Boneage (BA) was calculated according to the methods of Greulich and Pyle (GP) using manual readings between 1993-2008 (n=368), and automated BA estimation from 2008-2013 (n=378) . Target height was calculated as the sum of the mother's and father's heights (cm) minus 13 cm, divided by 2. Predicted Adult Height (PAH) was calculated using BoneXpert .

17β-Estradiol treatment

The decision to initiate treatment with E2 was determined individually, and made by the physician together with the patient and her parents, depending on height SDS, age, PAH and target height. Oral E2 was administered in increasing doses depending on age and pubertal stage. The starting doses ranged between 0.2 mg E2 to 4 mg E2. The speed of dose increment depended on the individual girl (age, bone BA, maturity, pubertal stage and PAH). The treatment consisted of 17β-estradiol supplemented with norethisteronacetat after 1-2 years of E2, or after the first menstrual bleeding. Oral E2 treatment was administered in the form of Trisekvens® (Novo Nordisk Scandinavia AB, Copenhagen, Denmark), Trisekvens Forte® (Novo Nordisk Scandinavia AB, Copenhagen, Denmark) and/or Femanest® (Sandoz A/S, Copenhagen, Denmark). Clinical and biochemical values were recorded at baseline and at each year thereafter. The treatment was generally terminated when the X-ray showed closed epiphyseal lines at final or near-final (<2 cm/year) height.

Laboratory analysis

Blood samples were drawn from the antecubital vein between 8 AM and 1 PM in the non-fasting state. Blood samples were clotted and centrifuged, and serum was stored at -20° Celsius until hormone analyses were performed. Serum follicle-stimulating hormone (FSH) and luteinising hormone (LH) were measured by time-resolved immunofluorometric assays (Delfia, Wallac, Turku, Finland). The detection limits (dL) for FSH and LH were 0.06 and 0.05 IU/l, respectively. Intra- and interassay coefficients of variation (CV) were < 5% in both gonadotropin assays. Testosterone was measured by radioimmunoassay (RIA) (Coat-a-count, Diagnostic Products Corporation, Los Angeles, CA) with a dL of 0.23 nmol/L and intra- and interassay CV both < 10%. Serum sex hormone-binding globulin (SHBG) was measured by time-resolved immunofluorometric assays (Delfia, Wallac, Turku, Finland) with a dL of 0.20 nmol/l, and intra- and interassay CVs of 5.8% and 6.4%, respectively. Serum insulin-like growth factor I (IGF-I) was measured using a highly sensitive in-house RIA as previously described by Juul et al. The intra- and interassay CV were 3.9% and 8.7%, respectively. From 2008 IGF-I levels were determined by conventional immunoassays (IMMULITE 2000 IGF-1; Siemens Healthcare Diagnostics, Los Angeles, CA, USA) on automated IMMULITE 2000 (Siemens). The CV were less than 4% and 9%, respectively. Serum insulin-like growth factor-binding protein 3 (IGFBP-3) was measured by RIA, as previously described by Blum et al. The intraassay CV was 2.4% and the interassay CV was 10.7%. Between 1993 and 2013, serum inhibin B was measured using one of two double antibody enzyme immunometric assays (Inhibin B DSL or Oxford Bio-Innovation Inhibin B), both with a dL of 20 pg/ml and intra- and interassay CV < 16%. Estradiol was measured by RIA (Pantex, Santa Monica, CA; before 1998 distributed by Immuno Diagnostic Systems, Bolton, UK) with a dL of 18 pmol/L, and intra- and interassay CVs < 8% and <13%, respectively. Only assays for IGF-I changed during the 20-year study period, and we compared the two assays rigorously and ensured that they yielded similar results before changing the assay.

Statistical analysis

Data are displayed as the median with interquartile range (25th;75th percentiles) and/or the range (min - max). Results of treatment effect and IGF-I (SD) are displayed as the mean ± SD. Hormone values below the dL of the assay were assigned a value corresponding to the dL/2. The Mann-Whitney U test and student's test was used to determine significance when comparing clinical, auxological, and laboratory data between groups, and student's t-test was used when comparing the effect of treatment within the group of girls treated with oral E2. All statistical analyses were performed using SPSS software (IBM Corporation, Armonk, NY, version 22).

ELIGIBILITY:
Inclusion Criteria:

* tall stature (height > 2 SD)

Exclusion Criteria:

* none

Ages: 1 Year to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients registered in our tertiary referral centre included
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
final height | 10 year observation time
  attainment of final height

CONTACTS AND LOCATIONS:
Overall Officials: Anders Juul, MD, Principal Investigator — Rigshospitalet, Denmark; Emmie Upners, student, Principal Investigator — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Upners EN, Juul A. Evaluation and phenotypic characteristics of 293 Danish girls with tall stature: effects of oral administration of natural 17beta-estradiol. Pediatr Res. 2016 Nov;80(5):693-701. doi: 10.1038/pr.2016.128. Epub 2016 Jun 20. PMID 27410906